CLINICAL TRIAL: NCT01889966
Title: Vasoreactivity Testing With Intravenous Sildenafil in Patients With Precapillary Pulmonary Hypertension (Treatment Optimisation Study)
Brief Title: VasoREACTivity Testing With Intravenous SILdenafil in Patients With Precapillary Pulmonary Hypertension
Acronym: SIL-REACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kerckhoff Heart Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dr. Andreas Rieth, Dr. med., senior physician cardiology, Kerckhoff Heart Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WS2196851
Record Dates: First submitted 2013-06-09; First posted 2013-07-01 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Pulmonary Hypertension Associated With Connective Tissue Disease
Keywords: vasoreactivity testing; Sildenafil; precapillary pulmonary hypertension; connective tissue disease; mean pressure in the pulmonary artery 25 mmHg or more; mean pulmonary capillary wedge pressure below 16 mmHg
MeSH Terms: conditions — Connective Tissue Diseases | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sildenafil (Experimental): oral Sildenafil 20 mg three times a day for 90 days
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — oral Sildenafil 3 x 20 mg for 90 days
  Other Names: Revatio; CAS15 number 139755-83-2; EV Substance code SUB10517MIG

SUMMARY:
Sildenafil is a selective pulmonary vasodilator; in patients with a special kind of pulmonary hypertension it is approved for treatment. The trial seeks to find out, whether the acute response to this treatment (= vasoreactivity testing) given intravenously is effective and allows prediction of therapy success during a following oral treatment.

ELIGIBILITY:
Inclusion Criteria:

* Precapillary pulmonary hypertension associated with connective tissue disease
* resting mean pressure in the pulmonary artery of > 24 mmHg
* resting mean pulmonary capillary wedge pressure (PCWP) of < 16 mmHg
* age 18 to 80 years
* women of childbearing potential must have a negative pregnancy test (ß-HCG in urine) and must use effective methods of contraception
* women must not be breastfeeding
* ability to understand and sign the informed consent, correctly signed informed consent

Exclusion Criteria:

* pretreatment with Sildenafil
* contraindications for Sildenafil treatment:

  * known intolerance to Sildenafil,
  * optic neuropathy (NAION),
  * known hereditary retina disease,
  * need of nitrate therapy
* advanced liver cirrhosis - CHILD C
* severely reduced renal function with GFR < 30 ml/min/1,73 m²
* stroke or myocardial infarction within the last 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
efficacy of Sildenafil I.V. for vasoreactivity testing | 1.5 hours
  Right heart catheterisation with comprehensive hemodynamic measurements (pressures in RA, RV, PA, PCW position; cardiac index (CI) by thermodilution; oxygen saturation in the PA; the same under exercise conditions) is performed. In case of precapillary pulmonary hypertension, Sildenafil is given I.V. and acute tolerability, safety and efficacy on hemodynamic parameters are registrated. Successful vasoreactivity testing is defined by lowering the mean PA pressure by 10 mmHg or more, lowering it below 40 mmHg and maintaining / rising of the CI. Safety is mainly defined by lack of a substantial effect of the study drug on systemic blood pressure.

SECONDARY OUTCOMES:
clinical efficacy of sildenafil per os predicted by testing it intravenously in the course of oral therapy | 90 days
  Complete hemodynamic and functional assessment after 90 days of oral Sildenafil therapy (same protocol as before except vasoreactivity testing). Hemodynamic parameters which characterize successful oral therapy are mainly mean PA-pressure (decrease), pulmonary vascular resistance (decrease) and cardiac index (increase) - at rest and exercise.
  Functional improvement is further characterized by exercise capacity (cardiopulmonary exercise testing: improvement of V´O2 peak by ≥ 1 ml/min/kg), fall of NTproBNP, improvement of echocardiographic parameters of right ventricular function (TAPSE, S´, RV-FAC).
  Evaluation, if positive initial vasoreactivity testing results in successful oral therapy as defined above.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas J Rieth, MD, Principal Investigator — Kerckhoff Heart Center
Locations (1):
- Kerckhoff Heart Center, Bad Nauheim, Germany

REFERENCES:
- [Derived] Rieth AJ, Richter MJ, Berkowitsch A, Frerix M, Tarner IH, Mitrovic V, Hamm CW. Intravenous sildenafil acutely improves hemodynamic response to exercise in patients with connective tissue disease. PLoS One. 2018 Sep 20;13(9):e0203947. doi: 10.1371/journal.pone.0203947. eCollection 2018. PMID 30235235